CLINICAL TRIAL: NCT03729609
Title: Drug Use Surveillance for ADCETRIS Intravenous Infusion "Untreated CD30-Positive Hodgkin's Lymphoma"
Brief Title: Drug Use Surveillance for Brentuximab Vedotin Intravenous Infusion "Untreated CD30-Positive Hodgkin's Lymphoma"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C25018; jRCT1080224121 (Registry Identifier: jRCT)
Record Dates: First submitted 2018-10-30; First posted 2018-11-02 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-03

CONDITIONS: Untreated CD30-Positive Hodgkin's Lymphoma
MeSH Terms: interventions — Brentuximab Vedotin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brentuximab vedotin 1.2 mg/kg (body weight): Brentuximab vedotin 1.2 milligrams per kilograms (mg/kg) (body weight), intravenous infusion, once every two weeks (up to 12 times). The dose should be adjusted depend on the participant's condition. Participants received interventions as part of routine medical care.
  Interventions: Drug: Brentuximab vedotin (Genetical Recombination)

INTERVENTIONS:
Drug: Brentuximab vedotin (Genetical Recombination) — Brentuximab vedotin Intravenous Infusion
  Other Names: ADCETRIS Intravenous Infusion 50 mg

SUMMARY:
The purpose of this survey is to monitor and identify the occurrence of neutropenia and febrile neutropenia in untreated CD30-positive Hodgkin's lymphoma participants on concomitant brentuximab vedotin and doxorubicin hydrochloride, vinblastine sulfate, and dacarbazine (AVD) in routine clinical practice.

DETAILED DESCRIPTION:
The drug being tested in this survey is called brentuximab vedotin intravenous infusion 50 mg. This intravenous infusion is being tested to treat people with untreated CD30-positive Hodgkin's lymphoma.

This survey is an observational (non-interventional) study and will look at the occurrence of neutropenia and febrile neutropenia in untreated CD30-positive Hodgkin's lymphoma patients on concomitant brentuximab vedotin and AVD in the routine clinical setting. The planned number of observed patients will be approximately 100.

This multi-center observational trial will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated participants
2. CD30-positive participants
3. Participants on concomitant Brentuximab vedotin and AVD

Exclusion Criteria:

1. Participants contraindicated for Brentuximab vedotin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with untreated CD30-positive Hodgkin's lymphoma on concomitant Brentuximab vedotin 1.2 mg/kg (body weight) and AVD as part of routine medical care.
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60214db2bf003ab495df

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 51 investigative sites in Japan, from 1 November 2018 to 27 September 2023.
Pre-assignment Details: Participants with a historical diagnosis of untreated CD30-Positive Hodgkin's lymphoma were enrolled. Participants received Brentuximab Vedotin Intravenous Infusion as part of a routine medical care.
Period: Overall Study
Arm/Group | Brentuximab Vedotin 1.2 mg/kg (Body Weight)
Started | 113
Completed | 112
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Brentuximab Vedotin 1.2 mg/kg (Body Weight)
Number analyzed (Participants) | 112
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.1 (19.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 112
Duration of Diagnosis of Hodgkin's Lymphoma [Mean (Standard Deviation); unit: Months] — Mean duration between the first diagnosis of Hodgkin's lymphoma and the first dose was reported. Population: The number analyzed is the number of participants with data available for analysis.
  Months
    number analyzed (Participants) | 111
    (all) | 2.3 (6.34)
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group performance status assess participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (greater than [>] 50 percent [%] of waking hours), capable of all self-care, unable to carry out any work activities; 3=capable of only limited selfcare, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed/chair; 5=dead.
  Participants
    Scale = 0 | 62
    Scale = 1 | 37
    Scale = 2 | 11
    Scale = 3 | 2
    Scale = 4 | 0
Healthcare Category [Count of Participants; unit: Participants]
  Outpatient | 2
  Inpatient | 110
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Medical Complications | 49
    Had Medical Complications | 63
Renal Impairment [Count of Participants; unit: Participants]
  Had No Renal Impairment | 109
  Had Renal Impairment | 3
Hepatic Impairment [Count of Participants; unit: Participants]
  Had No Hepatic Impairment | 109
  Had Hepatic Impairment | 3
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had No Medical History | 65
    Had Medical History | 47
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 58.26 (12.450)
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2]
  Kilogram (kg)/meter (m)^2 | 22.20 (3.561)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade 3 or Higher Neutropenia and Febrile Neutropenia
Description: Severity grades was evaluated as per National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE). Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life-threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to AE.
Time Frame: Up to 2 weeks after the last dose (approximately 6 months)
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin 1.2 mg/kg (Body Weight)
Number analyzed (Participants) | 112
Participants
  Neutropenia | 65
  Febrile Neutropenia | 31

2. Secondary Outcome: Tumor Response Rate Based on Investigator's Assessment
Description: Tumor response rate was defined as the percentage of participants with complete response (CR) or partial response (PR) as assessed by the Revised response criteria for malignant lymphoma by Cheson. CR is defined as the disappearance of all evidence of disease and PR is defined as regression of measurable disease and no new sites.
Time Frame: Baseline, Up to 2 weeks after the last dose (approximately 6 months)
Population: Efficacy analysis set: all participants who received at least one dose of protocol treatment without major protocol deviation. The number analyzed was the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin 1.2 mg/kg (Body Weight)
Number analyzed (Participants) | 98
Participants | 87

ADVERSE EVENTS:
Time Frame: Up to 2 weeks after the last dose (approximately 6 months)
Description: At each visit the investigator had to document any occurrence of Neutropenia and Febrile Neutropenia with Grade 3 or higher events as AEs, irrespective of the relation to the survey treatment. Only Neutropenia and Febrile Neutropenia with Grade 3 or higher events were planned to be collected and assessed in this study. The other AEs were out of the scope for the data collection plan.
Arm/Group | Brentuximab Vedotin 1.2 mg/kg (Body Weight)
All-Cause Mortality (participants affected / at risk) | 1/112
Serious Adverse Events (participants affected / at risk) | 44/112
Other Adverse Events (participants affected / at risk) | 52/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin 1.2 mg/kg (Body Weight) (N=112)
Febrile Neutropenia (Blood and lymphatic system disorders) | 31
Neutropenia (Investigations) | 13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin 1.2 mg/kg (Body Weight) (N=112)
Neutropenia (Investigations) | 52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT03729609/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT03729609/SAP_001.pdf